CLINICAL TRIAL: NCT03704207
Title: Utility of PCD Diagnostics to Improve Clinical Care
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Vanderbilt University Medical Center (Other)
Responsible Party: Principal Investigator, Michael O'Connor, Assistant Professor, Vanderbilt University Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: IRB #160951
Record Dates: First submitted 2018-10-08; First posted 2018-10-12 (Actual); Last update posted 2025-07-01 (Actual); Status verified 2025-06

CONDITIONS: Primary Ciliary Dyskinesia
MeSH Terms: conditions — Ciliary Motility Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Nasal Nitric Oxide testing and collection of clinical data (Other): Participants will have nNO testing is indicated. All participants in this study have some basic clinical data collected at time of enrollment. Participants with a confirmed diagnosis of PCD or in those participants with a working diagnosis of PCD in which ongoing nNO testing is performed have prospective data collection. Some participants have a confirmed diagnosis of PCD by genetics or ciliary biopsy at time of study entry and thus do not need nNO testing, but are followed prospectively with collection of basic clinical data
  Interventions: Other: nNO testing

INTERVENTIONS:
Other: nNO testing — Collection of already performed clinical data and nNO testing

SUMMARY:
This is a study evaluating the utility of current Primary Ciliary Dyskinesia (PCD) diagnostic tests, including nasal nitric oxide testing.

DETAILED DESCRIPTION:
This study is a prospective data collection of individuals referred to the investigators clinical center for considerations of PCD. Participants sign informed consent to have clinical information entered into a secure electronic database. As part of this study, participants may have nasal nitric oxide (nNO) testing performed. nNO testing is a research procedure, but it is a test with growing utility for making a diagnosis of PCD when performed in the right clinical setting.

ELIGIBILITY:
Inclusion Criteria:

* Referred to center for PCD diagnosis considerations
* Ability to perform study procedures
* Age greater than 2 years of age

Exclusion Criteria:

* Age less than 2 years of age Inability to perform informed consent

Min Age: 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2017-06-01 (Actual); Primary Completion 2028-06-01 (Estimated); Study Completion 2028-06-01 (Estimated)

PRIMARY OUTCOMES:
frequency of nNO tests performed | 3 years
  number of tests
Frequency of genetic tests performed | 3 years
  number of tests

CONTACTS AND LOCATIONS:
Locations (1):
- Vanderbilt Children's hospital, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No